CLINICAL TRIAL: NCT01787006
Title: Definitive Radiochemotherapy With 5-FU / Cisplatin Plus/Minus Cetuximab in Unresectable Locally Advanced Esophageal Cancer: a Phase II Study
Brief Title: Definitive Radiochemotherapy Plus/Minus Cetuximab in Unresectable Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dirk Rades, MD, Professor Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEOPARD II; 2010-023427-18 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Cancer
Keywords: non resectable; locally advanced; Cetuximab; radiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cetuximab; Cisplatin; Fluorouracil; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab, Cisplatin, 5-FU, Radiotherapy (Experimental): Cetuximab: Initial doses 400mg/m2 (day 1), followed by weekly doses of 250mg/m2 for 14 weeks in total, IV
  5-fluorouracil (5-FU): 1000mg/m2 per day as continuous infusion on day 8-11 and 36-39, 750mg/m2/day as continuous infusion on day 71-74 and 99-102
  Cisplatin 20mg/m2/day as intravenous bolus over 60 min on day 1-4 of every cycle (day 8-11, 36-39, 71-74 and 99-102)
  radiotherapy: 59.4 Gy (33 fractions of 1.8 Gy) over 6.5-7 weeks (5 x 1.8 Gy per week)on primary tumor. 50.4 Gy on locoregional lymphnodes. If resectability is reached after 4-4.5 weeks (36-41.4 Gy) the radiotherapy stops after 45 Gy and the patient undergoes surgery.
  Interventions: Drug: Cetuximab; Drug: Cisplatin, 5-FU; Radiation: Radiotherapy
- Cisplatin, 5-FU, Radiotherapy (Active Comparator): 5-FU: 1000mg/m2 per day as continuous infusion on day 1-4 and 29-32, 750mg/m2/day as continuous infusion on day 64-67 and 92-95
  Cisplatin 20mg/m2/day as intravenous bolus over 60 min on day 1-4 of every cycle (day 1-4, 29-32, 64-67 and 92-95)
  radiotherapy: 59.4 Gy (33 fractions of 1.8 Gy) over 6.5-7 weeks (5 x 1.8 Gy per week)on primary tumor. 50.4 Gy on locoregional lymphnodes. If resectability is reached after 4-4.5 weeks (36-41.4 Gy) the radiotherapy stops after 45 Gy and the patient undergoes surgery.
  Interventions: Drug: Cisplatin, 5-FU; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — Initial doses 400mg/m2 (day 1), followed by weekly doses of 250mg/m2 for 14 weeks in total
  Other Names: Erbitux
  Arms: Cetuximab, Cisplatin, 5-FU, Radiotherapy
Drug: Cisplatin, 5-FU — 5-FU: 1000mg/m2 per day as continuous infusion on day 1-4 of cycle 1 and 2, 750mg/m2/day as continuous infusion on day 1-4 of cycle 3 and 4
  Cisplatin 20mg/m2/day as intravenous bolus over 60 min on day 1-4 of every cycle
  Other Names: CDDP, 5-fluorouracil
Radiation: Radiotherapy — 59.4 Gy (33 fractions of 1.8 Gy) over 6.5-7 weeks (5 x 1.8 Gy per week)on primary tumor. 50.4 Gy on locoregional lymphnodes. If resectability is reached after 4-4.5 weeks (36-41.4 Gy) the radiotherapy stops after 45 Gy and the patient undergoes surgery.
  Other Names: Irradiation

SUMMARY:
Esophageal cancer is a highly aggressive tumor. Treatment options are various and range from chemotherapy to radiotherapy and several surgical techniques. Nevertheless, the overall survival rates for this disease remain poor.

During the last years the combination of cetuximab with standard chemotherapy or radiotherapy has mainly be investigated in clinical trials focusing on colorectal and/or head and neck cancer.

The results obtained from theses studies were very encouraging and led to the initiation of active clinical research in esophageal cancer patients with antibody inhibition of the epidermal growth factor receptor (EGFR).

The first data in this indication are encouraging showing that cetuximab can safely be added to chemoradiation for esophageal cancer patients with first hints of efficacy.

Based on the experiences with cetuximab in colorectal cancer and in combination with radiotherapy in head and neck cancer, the aim of the present study is to evaluate the feasibility of a combined treatment of cetuximab with continuous infusional 5-FU, cisplatin and radiotherapy in patients with esophageal cancer and to assess if the overall survival rates can be increased by addition of an EGFR-targeted therapy.

DETAILED DESCRIPTION:
Esophageal cancer is a highly aggressive neoplasm which is fatal in the great majority of patients. On a global basis, cancer of the esophagus is the sixth leading cause of cancer death worldwide. In fact, gastric and esophageal cancers together accounted for nearly 1.3 million new cases and 980,000 deaths worldwide in 2000 - more than lung, breast, or colorectal cancer. With advances in surgical techniques and treatment, the prognosis of esophageal cancer has slowly improved over the past decades. However, with a 5-year overall survival rate of approximately 14%, at the time of development of the LEOPARD-II protocol, survival was poor, even in comparison with the dismal survival rates (4%) from the 1970s. Underlying reasons for this disappointingly low survival rate are above all the difficulties in cancer detection at an advanced stage, with over 50% of patients with unresectable disease or distant metastasis at presentation and the limited survival achieved with palliative chemotherapy alone for patients with metastatic or unresectable disease.

Clearly, additional strategies are needed to improve the systemic treatment options for esophageal cancer.

The optimal treatment of locally advanced esophageal cancer, a potentially curable disease, is controversial. Through several non-randomized cooperative group trials, concurrent cisplatin-based chemoradiation or surgery alone represent acceptable standards of care for patients with resectable tumors.

Metastatic or unresectable esophageal cancer is found at presentation in more than 50% of patients and is considered incurable. At the time of protocol development, chemotherapy was palliative, improving quality of life and dysphagia in 60%-80% of patients. Typical clinical and radiographic responses lasted for fewer than 4 months, with a median overall survival time of 8-10 months.

Combination chemotherapies have been demonstrated to be superior to best supportive care and chemotherapy given as a single agent, with occasional patients achieving complete responses (0%-11%). However, even with the combination regimens, the median survival time remained less than 10 months.

An improved understanding of the molecular pathogenesis of cancer has facilitated the development of novel agents designed to target critical pathways involved in cancer development and progression. Epidermal growth factor receptor (EGFR) plays a crucial role in tumour growth. EGFR-dependent signaling is involved in cell proliferation, apoptosis, angiogenesis, and metastatic spread.

The overexpression of EGFR has repeatedly been shown to predict poor prognosis in both esophageal squamous cell carcinoma and gastro esophageal junction adenocarcinoma. EGFR blockade through monoclonal antibodies (Cetuximab, Matuzumab and Panitumumab) and tyrosine kinase inhibitors (gefitinib, erlotinib) has translated into promising evidence of clinical benefit in clinical trials.

Cetuximab is a targeted therapeutic agent, a chimeric monoclonal antibody that specifically binds to the EGFR with high affinity, internalising the receptor and preventing ligands from interacting with the receptors and thus effectively blocking ligand-induced EGFR phosphorylation. In addition, cetuximab had been found to potentiate the effects of chemotherapy and radiotherapy in experimental systems. The dose of cetuximab (initial dose 400 mg/m2 and subsequent weekly doses of 250 mg/m2) has been found to be generally safe and effective in several studies in major tumor types expressing the EGFR. These included colorectal cancer and squamous cell carcinoma of the head and neck, with cetuximab given either in combination studies with chemotherapy and radiotherapy or as monotherapy.

In two phase I studies prior to LEOPARD-II, EGFR-directed antibodies had shown activity in patients with esophageal cancer. In the phase I study of the humanized EGFR monoclonal antibody (mAb) EMD72000, one patient with metastatic, pretreated squamous cell carcinoma had had a durable, 6-month partial response.

In addition, a phase I trial with a fully human EGFR mAb, had reported stable disease for 7 months in one esophageal cancer patient. Preclinical and these early clinical studies suggested potential activity and minimal toxicities with EGFR antibodies for esophageal cancer.

Furthermore, a randomised phase II compared cisplatin + 5-FU (CF) to cisplatin + 5-FU + cetuximab (CET-CF) (n=62). Cetuximab did not increase grade 3/4 toxicity, except for rash (6% versus 0%) and diarrhea (16% versus 0%). The overall response rates were 19% and 13% for the CET-CF and CF arms respectively, and the disease control rates were 75% and 57%, respectively. The median progression free survival was 5.9 and 3.6 months and median overall survival 9.5 and 5.5 months for CET-CF and CF, respectively.

With respect to the combination of Cetuximab with radiotherapy, preclinical studies have shown, that Cetuximab enhanced the radiosensitivity of EGFR expressing tumour cells in vitro and in tumour xenografts and the repopulation of epithelial tumour cells after exposure to radiation was related to the activation and expression of EGFR. Cetuximab also enhanced the efficacy of docetaxel chemoradiotherapy in human adenocarcinoma xenografts.

Rationale for the LEOPARD-II study Esophageal cancer is a highly aggressive tumor and one of the most frequent malignant diseases worldwide.

Treatment options are various and range from chemotherapy to radiotherapy and several surgical techniques. Nevertheless, the overall survival rates for this disease remain poor. During the last years before protocol development the combination of cetuximab with standard chemotherapy or radiotherapy had mainly been investigated in clinical trials focusing on colorectal and/or head and neck cancer. The results obtained from these studies had been very encouraging and led to the initiation of active clinical research in esophageal cancer patients with antibody inhibition of the EGFR. The first data in this indication were encouraging showing that cetuximab could safely be added to chemoradiation for esophageal cancer patients with first hints of efficacy. Based on the experiences with cetuximab in colorectal cancer and in combination with radiotherapy in head and neck cancer, the aim of the LEOPARD-II study was to evaluate the feasibility of a combined treatment of cetuximab with continuous infusional 5-FU, cisplatin and radiotherapy in patients with esophageal cancer and to assess if the overall survival rates could be increased by addition of an EGFR-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Dated and signed written informed consent
* Male or female patients between 18 years and 75 years; patients > 75 years if their karnofsky performance status is ≥ 80.
* Histologically proven squamous cell carcinoma or adenocarcinoma of the esophagus which is not curatively resectable. Resectability has to be defined by a surgeon before radiochemotherapy. The tumor is considered unresectable due to T-stage, N-stage, performance status, nutritional status, co-morbidity (pulmonal function, other), tumor location upper third or other reasons
* Karnofsky Performance Status ≥ 70
* Women of child-bearing potential must have a negative pregnancy test
* Adequate cardial-, pulmonal- and ear function

Adequate bone marrow function:

* leukocytes ≥ 3.0 x 10^9/L
* neutrophiles ≥ 1.5 x 10^9/L
* thrombocytes ≥ 100 x 10^9/L
* hemoglobin ≥ 10.0 g/dl

Adequate liver function:

* bilirubin ≤ 2.0 mg/dl
* transaminases (serum glutamic pyruvic transaminase (SGPT), serum glutamic oxaloacetic transaminase (SGOT), gamma-GT) ≤ 3 x upper limit of normal (ULN)

Adequate kidney function:

* serum creatinine ≤ 1.5 mg/dl
* creatinine clearance ≥ 50 ml/min according to Cockcroft-Gault Formula
* no known allergies against chimeric antibodies
* effective contraception for male and female patients if there is a risk of conception

Exclusion Criteria:

* distant metastasis
* previous treatment of esophageal cancer
* previous therapy with monoclonal antibodies and / or EGFR-targeted therapy
* previous second malignancies with exception of a history of a previous curatively treated basal cell carcinoma of the skin or pre-invasive cervix carcinoma
* serious concomitant disease or medical condition
* lung function: forced expiratory volume in one second (FEV1)) < 1.1
* clinically relevant coronary artery diseases or known myocardial infarction within the last 12 months or ventricular ejection fraction (LVEF) below normal
* every active dermatological condition > grade 1
* contraindications to receive cisplatin, 5-FU or cetuximab
* concurrent treatment with other experimental drugs or participation in another clinical trial within 30 days before study start
* patient pregnant or breast feeding
* known drug abuse, medication abuse, alcohol abuse
* social situations limiting the compliance with the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-09; Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr., Principal Investigator — Universität zu Lübeck, Klinik für Strahlentherapie
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Klinik für Strahlentherapie, Lübeck, Germany

REFERENCES:
- [Derived] Rades D, Bartscht T, Hunold P, Schmidberger H, Konig L, Debus J, Belka C, Homann N, Spillner P, Petersen C, Kuhnt T, Fietkau R, Ridwelski K, Karcher-Kilian K, Kranich A, Mannikko S, Schild SE, Maderer A, Moehler M. Radiochemotherapy with or without cetuximab for unresectable esophageal cancer: final results of a randomized phase 2 trial (LEOPARD-2). Strahlenther Onkol. 2020 Sep;196(9):795-804. doi: 10.1007/s00066-020-01646-4. Epub 2020 Jun 12. PMID 32533228

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab, Cisplatin, 5-FU, Radiotherapy: Cetuximab: Initial doses 400mg/m2 (day 1), followed by weekly doses of 250mg/m2 for 14 weeks in total, IV
  5-FU: 1000mg/m2 per day as continuous infusion on day 8-11 and 36-39, 750mg/m2/day as continuous infusion on day 71-74 and 99-102
  Cisplatin 20mg/m2/day as intravenous bolus over 60 min on day 1-4 of every cycle (day 8-11, 36-39, 71-74 and 99-102)
  radiotherapy: 59.4 Gy (33 fractions of 1.8 Gy) over 6.5-7 weeks (5 x 1.8 Gy per week)on primary tumor. 50.4 Gy on locoregional lymphnodes. If resectability is reached after 4-4.5 weeks (36-41.4 Gy) the radiotherapy stops after 45 Gy and the patient undergoes surgery.
Period: Overall Study
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Started | 35 | 39
Completed | 32 | 36
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Median (Full Range); unit: years]
  median | 65 [44 to 80] | 64 [49 to 79] | 65 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 22 | 30 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic origin: Caucasian | 32 | 36 | 68
  Ethnic origin: Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 32 | 36 | 68
Histology [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 27 | 28 | 55
  Adeno carcinoma | 5 | 8 | 13
Histologic grading [Count of Participants; unit: Participants] — The histological grading was performed using the following scale:
  GX Grade cannot be assessed G1 Well differentiated (Low grade) G2 Moderately differentiated (Intermediate grade) G3 Poorly differentiated (High grade)
  Participants
    G1 | 0 | 1 | 1
    G2 | 16 | 18 | 34
    G3 | 11 | 10 | 21
    Gx | 5 | 7 | 12
clinical T-category [Count of Participants; unit: Participants] — T describes the size depth of local invasion by the primary tumor. A higher T-category represents a more advanced primary tumor, generally associated with a worse prognosis. Patients were staged for T-category using computed tomography and endoscopic ultrasound.
  Participants
    cT1 | 1 | 1 | 2
    cT2 | 2 | 0 | 2
    cT3 | 20 | 20 | 40
    cT4 | 8 | 13 | 21
    cTx | 1 | 2 | 3
clinical N-category [Count of Participants; unit: Participants] — N describes the extent of the involvement of regional lymph nodes. A higher N-category represents a higher number of refional lymph nodes, generally associated with a worse prognosis. Patients were staged for N-category using computed tomography and endoscopic ultrasound.
  Participants
    cN0 | 7 | 8 | 15
    cN1 | 14 | 14 | 28
    cN2 | 7 | 7 | 14
    cN3 | 3 | 3 | 6
    cNx | 0 | 3 | 3
    cN+ | 1 | 1 | 2
clinical M-category [Count of Participants; unit: Participants] — M describes thew presence or absence of distant metastasis. In the 6th edition of the TNM-classification, M1a indicated metastases to the cervical or celiac axis lymph nodes, and M1b metastases to distant sites. The TNM-classification from 2009 (7th edition) used only M0 (absence) and M1 (presence) for distant metastasis. M1 is generally associated with a worse prognosis. Patients were staged for M-category using computed tomography (thorax and abdomen).
  Participants
    cM0 | 31 | 35 | 66
    cM1 (formerly cM1a) | 0 | 1 | 1
    cMx | 1 | 0 | 1
Tumor site [Count of Participants; unit: Participants]
  Lower third only | 9 | 15 | 24
  Lower and middle third | 1 | 3 | 4
  Middle third only | 13 | 8 | 21
  Upper and middle third | 0 | 2 | 2
  Upper third only | 9 | 6 | 15
  Not specified | 0 | 2 | 2
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — 100 - Normal; no evidence of disease. 90 - Normal activity; minor signs/symptoms. 80 - Normal activity with effort; some signs/symptoms. 70 - Cares for self; unable for normal activity or active work. 60 - Requires occasional assistance, cares for most personal needs. 50 - Requires considerable assistance + frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospital admission indicated. 20 - Very sick; hospital admission + supportive treatment necessary. 10 - Moribund; fatal processes progressing rapidly. 0 - Dead
  Participants
    KPS of 70 | 1 | 2 | 3
    KPS of 80-100 | 31 | 34 | 65

OUTCOME MEASURES:

1. Primary Outcome: Rate of Participants Who Were Alive at 2 Years
Description: Overall Survival (OS) was defined as freedom from death of any cause. Time to death was calculated from the day of randomization, and the patients were followed for a maximum of 24 months (2 years).
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 71 [55 to 87] | 53 [36 to 71]

2. Secondary Outcome: Rate of Participants Who Were Alive at 1 Year
Description: Overall Survival (OS) was defined as freedom from death of any cause. Time to death was calculated from the day of randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 74 [59 to 90] | 70 [54 to 86]

3. Secondary Outcome: Rate of Participants Who Were Alive Without Progression of Disease at 1 Year
Description: For progression-free survival (PFS), the event was defined as first occurrence of radiologically proven progression or clinical progression or death due to progressive disease. Time to event was referenced from the day of randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 64 [47 to 82] | 58 [40 to 75]

4. Secondary Outcome: Rate of Participants Who Were Alive Without Progression of Disease at 2 Years
Description: as for outcome 3
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 56 [37 to 75] | 44 [26 to 62]

5. Secondary Outcome: Number of Participants Experiencing at Least One Grade >=3 Toxicity
Description: Toxicity was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) (version 4.03).
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
Participants
  at least one grade >=3 toxicity | 26 | 27
  no grade >=3 toxicity | 6 | 9

6. Secondary Outcome: Rate of Participants Who Were Alive Without Distant Metastases at 1 Year
Description: For metastases-free survival (MFS), the event was defined as first occurrence of distant metastasis. Time to event was referenced from the day of randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 79 [64 to 94] | 70 [53 to 86]

7. Secondary Outcome: Rate of Participants Who Were Alive Without Distant Metastases at 2 Years
Description: as for outcome 6
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 74 [57 to 91] | 54 [36 to 73]

8. Secondary Outcome: Number of Participants Who Achieved at Least Partial Response (Responders)
Description: Response was defined according to the RECIST criteria (Version 1.1) based on the assessments (computed tomography, magnetic resonance imaging or other) for target lesions, non-target lesions as well as considering the occurrence of new lesions.
  The best overall response (RECIST) was chosen for each patient out of all valid tumour assessments before start of next-line therapy (complete response=CR being the best and progressive disease=PD the worst). Frequencies with percentages were to be given for each category (CR, partial response (PR), stable disease (SD), PD) by treatment group. The data were to be presented as the dichotomous endpoint of objective response, for which patients with best overall response of CR or PR were considered as responders, and those with best overall response of SD or PD as non-responders. The difference between objective response rates in the two treatment arms was to be compared with a Chi-square test.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
Participants
  responders | 26 | 25
  non-responders | 6 | 11

9. Secondary Outcome: Rate of Participants Who Were Alive Without Loco-regional Failure at 1 Year
Description: Loco-regional failure was defined as progressive primary tumor and/or regional lymph nodes on endoscopy, endoscopic ultrasound or computed tomography.Time to event was referenced from the day of randomization.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 89 [77 to 100] | 81 [67 to 95]

10. Secondary Outcome: Rate of Participants Who Were Alive Without Loco-regional Failure at 2 Years
Description: Loco-regional failure was defined as progressive primary tumor and/or regional lymph nodes on endoscopy, endoscopic ultrasound or computed tomography. Time to event was referenced from the day of randomization.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 32 | 36
percentage of participants | 84 [70 to 99] | 72 [55 to 89]

11. Secondary Outcome: Change in Quality of Life Between Baseline and End of Treatment (After 5 to 13 Weeks)
Description: Quality of Life was assessed with EORTC QLQ-C30 and QLQ-OES18 questionnaires. For QLQ-C30, global health status, functional scales (physical, role, emotional, cognitive and social functioning) and symptom scales (fatigue, nausea/vomiting, pain, dyspnea, loss of appetite, constipation, diarrhea, financial difficulties) were calculated. Scores ranged from 0 to 100; higher scores represented higher levels of quality of life, functioning, or symptoms/problems. Score were calculated using mean values.
  For QLQ-OES18, symptom scales (problems with eating, reflux, pain, problems swallowing saliva, dry mouth, taste disorders, problems while coughing or speaking) and functional scale (dysphagia) were assessed the same way.
  A change between two time points, i.e. baseline (prior to treatment) and end of treatment (after 5 to 13 weeks, depending on treatment arm (6.5 weeks without and 13 weeks with cetuximab) and achievement of resectability (end of treatment after 5 weeks), is reported.
Time Frame: end of treatment (after 5 to 13 weeks)
Population: All scales used for the rows below in the outcome measure data table ranged between 0 and 100.
  For scales indicated [H], a higher score represents a better situation (quality of life, functioning).
  For scales indicated [L], a lower value represents a better outcome (symptoms/problems).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
Number analyzed (Participants) | 23 | 26
score on a scale
  Change in global health status [H] | -9.1 (23.96) | -4.7 (33.41)
  Change in physical functioning [H] | -19.2 (27.34) | -13.0 (24.66)
  Change in role functioning [H] | -22.0 (32.69) | -18.1 (28.39)
  Change in emotional functioning [H] | -9.4 (25.54) | 3.4 (27.52)
  Change in cognitive functioning [H] | -13.8 (24.95) | -7.2 (21.80)
  Change in social functioning [H] | -12.1 (37.86) | -3.6 (42.03)
  Change regarding fatigue [L] | 21.7 (24.50) | 15.5 (33.92)
  Change regarding nausea/vomiting [L] | 23.2 (30.46) | 21.7 (29.06)
  Change regarding pain [L] | -2.2 (27.66) | 2.1 (37.85)
  Change regarding dyspnoea [L] | 10.1 (23.43) | 11.6 (39.71)
  Change regarding insomnia [L] | -10.1 (35.44) | 14.5 (41.23)
  Change regarding loss of appetite [L] | 23.2 (43.15) | 31.9 (50.73)
  Change regarding constipation [L] | 13.0 (29.71) | -1.4 (39.54)
  Change regarding diarrhea [L] | 15.2 (24.62) | 2.9 (19.88)
  Change regarding financial difficulties [L] | 0.0 (36.24) | -5.8 (38.47)
  Change regarding problems with eating [L] | 4.0 (34.07) | 1.9 (36.20)
  Change regarding reflux [L] | 11.6 (28.62) | -1.4 (35.86)
  Change regarding pain while eating [L] | 2.9 (18.42) | -6.5 (35.24)
  Change regarding problems swallowing saliva [L] | -2.9 (41.33) | 4.3 (30.66)
  Change regarding dry mouth [L] | 21.7 (38.41) | 1.5 (41.76)
  Change regarding taste disorders [L] | 33.3 (46.06) | 27.3 (39.36)
  Change regarding problems while coughing [L] | -1.4 (34.05) | 15.9 (28.19)
  Dysphagia [H] | -10.1 (33.41) | 0.0 (35.93)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Common Terminology Criteria for Adverse Events (CTCAE), version 4.03
Arm/Group | Cetuximab, Cisplatin, 5-FU, Radiotherapy | Cisplatin, 5-FU, Radiotherapy
All-Cause Mortality (participants affected / at risk) | 13/32 | 20/36
Serious Adverse Events (participants affected / at risk) | 21/32 | 24/36
Other Adverse Events (participants affected / at risk) | 32/32 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Cisplatin, 5-FU, Radiotherapy (N=32) | Cisplatin, 5-FU, Radiotherapy (N=36)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (11)
Esophagitis (Gastrointestinal disorders) | 6 (7) | 5 (5)
White blood cell decreased (Investigations) | 3 (3) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5)
Hypokalemia (low potassium) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Stoma site infection (Infections and infestations) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Liver enzymes increased/elevated (Investigations) | 1 (1) | 3 (3)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Infection (not specified) (Infections and infestations) | 2 (2) | 1 (1)
Pancytopenia (Investigations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (not specified) (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Immune system disorder (not specified) (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocilitis (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Morphine overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tumor bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Doslocation of feeding tube (PEG) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration/Exsiccosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 2 (2) | 2 (3)
Nephrotoxicity, tubular function impaired (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palma-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Acneiforme rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reduced overall health condition (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab, Cisplatin, 5-FU, Radiotherapy (N=32) | Cisplatin, 5-FU, Radiotherapy (N=36)
Nausea (Gastrointestinal disorders) | 19 | 20
Hypokalemia (low potassium) (Metabolism and nutrition disorders) | 16 | 12
Anemia (Blood and lymphatic system disorders) | 13 | 13
Fatigue (General disorders) | 9 | 18
Esophagitis (Gastrointestinal disorders) | 11 | 14
White blood cell decreased (Investigations) | 16 | 8
Dysphagia (Gastrointestinal disorders) | 9 | 9
Platelet count decreased (Investigations) | 11 | 7
Constipation (Gastrointestinal disorders) | 6 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 13 | 3
Vomiting (Gastrointestinal disorders) | 6 | 7
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Diarrhea (Gastrointestinal disorders) | 7 | 5
Oral mucositis (Gastrointestinal disorders) | 8 | 4
Weight loss (General disorders) | 9 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 2
Acneiforme rash (Skin and subcutaneous tissue disorders) | 11 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 9 | 1
Edema (General disorders) | 6 | 4
Neutrophil count decreased (Investigations) | 5 | 4
Dizziness (Nervous system disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Maculopapular rash (Skin and subcutaneous tissue disorders) | 7 | 1
Pain (General disorders) | 5 | 2
Insomnia (Nervous system disorders) | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
GGT increased (Investigations) | 3 | 3
Infection (not specified) (Infections and infestations) | 3 | 2
Paresthesia (Nervous system disorders) | 1 | 4
Thrombembolic event (Vascular disorders) | 2 | 3
Allergic reaction (Immune system disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Stoma site infection (Infections and infestations) | 3 | 1
Hyponatremia (low sodium) (Metabolism and nutrition disorders) | 1 | 3
Weight gain (General disorders) | 0 | 4
Syncope (Nervous system disorders) | 2 | 2
Urinary retention (Renal and urinary disorders) | 2 | 2
Esophageal pain (Gastrointestinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications (presentation of results obtained at a participating center at scientific meetings or publication of these results) prior to public release and can embargo communications regarding trial results prior to submission of the results of the entire study for publication.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01787006/Prot_SAP_000.pdf
  • Informed Consent Form (2012-08-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01787006/ICF_001.pdf